CLINICAL TRIAL: NCT05148260
Title: Tackling Postnatal Depression: Culturally Adapted Learning Through Play Plus (LTP+) Intervention for Depressed British Mothers of African and Caribbean Origin
Brief Title: Tackling Postnatal Depression: Culturally Adapted Learning Through Play Plus (LTP+) Intervention for British Mothers of African and Caribbean Origin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Dr Dung Jidong, PhD, Senior Lecturer, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-0001-5034-0335b
Record Dates: First submitted 2021-11-11; First posted 2021-12-08 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Postnatal Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Long-Term Potentiation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP+ (Experimental): The LTP+ is divided into two components:
  First, underpinned by Piaget's theory of cognitive development (Piaget, 1952; Sidik, 2020) and Bowlby's theory of attachment (Bowlby, 1980; Granqvist & Duschinsky, 2021), the central focus here is a pictorial calendar devised for parents, depicting eight successive stages of child development from birth to 3 years, with illustrations of parent-child play and other activities that promote parental involvement, learning, and mum-baby attachment.
  Second, well-grounded in the standard framework of cognitive-behavioural theory (Bernal et al., 2009) and uses techniques of active listening, changing negative thinking, guided discovery, behavioural tasks, and homework (i.e. trying things out between sessions, putting what has been learnt into practice), while educating participating mums about depression/anxiety, correlates and management, social support, and practical advice on using appropriate healthcare (Bernal et al., 2009).
  Interventions: Behavioral: Learning Through Play plus (LTP+)
- Psychoeducation (Active Comparator): This is the comparative group with a primary aim of monitoring participating mums to ensure their postnatal depression does not degenerate. However, supportive, and postnatal educational components are provided. These psychoeducation sessions are grounded on the theory and philosophy of group psychosocial support (with basic but relevant topics on postnatal mental healthcare advice and discussions).
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Learning Through Play plus (LTP+) — Group-1: Experimental (n=40 participants) will receive the LTP+ which consist of a total of 12-group integrated treatment sessions lasting approximately 60-90 minutes per session every fortnight with 10 mother/child pair per sub-group.
  Arms: LTP+
Behavioral: Psychoeducation — Group-2: Controlled (n=40 participants) will receive 'psychoeducation' which consist of a total of 12-group sessions lasting approximately 60-90 minutes per session every fortnight with 10 mother-child pair per sub-group.
  Arms: Psychoeducation

SUMMARY:
By 2030, depression will be the leading global disease burden. Postnatal depression due to childbirth/parenting leads to long-term negative consequences for mothers, their children and their families. The British African/Caribbean communities are worse hit by the unprecedented impact of post-Covid-19-syndromes, leading to an exponential increase in postnatal depression. Yet, the uptake of mental healthcare by British mothers of African and Caribbean origin is low due to limited access to culturally appropriate care. Theories of attachment and cognitivism were innovatively integrated to examine Learning-Through-Play plus (LTP+) intervention for postnatal depression using a pilot randomised controlled trial. The proposed LTP+ is co-developed and ecologically friendly because it is manualised and can be delivered by non-mental health specialists such as trained community health workers who are more culturally knowledgeable. Findings will be disseminated through academic publications/presentations, policy briefs, original animated videos and podcast series laying the foundations for a psychosocial approach to tackling postnatal depression

ELIGIBILITY:
Inclusion Criteria

Only British mothers of African and Caribbean heritage:

* experiencing emotional distress due to childbirth or parenting and scored 5 or above on the patient health questionnaire (PHQ-9)
* who have children age 0-3 years
* residents of designated communities and available for follow-up
* are 18 years and above
* able to give informed consent.

Exclusion Criteria

Are mothers:

* with a medical condition that would prevent their participation such as active suicidal ideation, tuberculosis, or heart failure
* temporary residents are unlikely to be available for follow up
* who are less than 18 years
* unable to provide consent.
* with non-British African and Caribbean heritage.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in postnatal depression is being assessed | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Primary outcome measure would be assessed using the Patient Health Questionnaire (PHQ-9)
Change in postnatal anxiety is being assessed | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Primary outcome measure would be assessed using the Generalised Anxiety Disorder (GAD7) scale
Change in social support is being assessed | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Primary outcome measures would be assessed using the Oslo Social Support Scale
Change in health-related quality of life is being assessed | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Outcome measure would be assessed using the Health-related Quality of Life scale (EuroQoL-5 Dimensions)
Change in service satisfaction is being assessed | Change is being assessed at 12 weeks end of intervention
  Outcome measure would be assessed using the brief Verona Service Satisfaction Scale
Change in child physio-emotional development is being assessed | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Outcome measure would be assessed using the Ages and Stages Social-Emotional Questionnaire
Change in parenting knowledge of child development is being assessed | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Outcome measure would be assessed using Learning Through Play Knowledge, Attitude and Practices (KAP) Questionnaire

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol